CLINICAL TRIAL: NCT04796714
Title: AntiPlatelet theraPy stratEgy followiNg Left Atrial appenDAGe closurE
Acronym: APPENDAGE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/29
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation; Atrial Appendage; Anticoagulants; Stroke; Platelet Aggregation Inhibitors
Keywords: left atrial appendage; percutaneous closure; stroke; antiplatelet therapy; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double antiplatelet therapy group (Sham Comparator): Patient randomized in this group will receive 1 tablet containing clopidogrel 75 mg and 1 bag containing aspirin 160 mg as treatment. This treatment will start on the day of LAAC procedure and continued for 3 months.
  Interventions: Drug: Double antiplatelet therapy; Device: Brain MRI; Other: Neurological tests
- Aspirin group (Experimental): Patients randomized in this group: will receive 1 bag containing aspirin 160 mg as treatment. This treatment will start on the day of LAAC procedure and continued for 3 months.
  Interventions: Drug: Aspirin; Device: Brain MRI; Other: Neurological tests

INTERVENTIONS:
Drug: Double antiplatelet therapy — One sachet of aspirin 160 mg and one tablet of clopidogrel 75 mg per day.during 3 months
  Arms: Double antiplatelet therapy group
Drug: Aspirin — One sachet of aspirin 160 mg per day during 3 months
  Arms: Aspirin group
Device: Brain MRI — Two cerebral Magnetic Resonance Imaging (MRI) examinations will be carried out (D0 and D90).
Other: Neurological tests — Neurological assessment with the implementation of the modified rankin, National Institute of Health Stroke Score (NIHSS), and Montreal Cognitive Assessment (MoCA) tests (D1 and M3)

SUMMARY:
The APPENDAGE study is a phase 4 multicentre randomized opened clinical trial comparing 2 different antithrombotic strategies following left atrial appendage closure (LAAC) in patients with non valvular atrial fibrillation (AF). The primary objective of the study is to evaluate the efficacy of Aspirin versus Aspirin + Clopidogrel after LAAC by comparing the occurrence of ischemic lesions on cerebrovascular magnetic resonance imaging (MRI) studies.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia and increases the risk of ischemic stroke. Although oral anticoagulation (OAC) is recommended in patients with CHADS2VA2SC score ≥ 1, this medication is associated with severe haemorrhagic complications. Several trials showed that percutaneous LAAC with the Watchman device (Boston Scientific, Natick, Massachusetts) or the Amplatzer Cardiac Plug (ACP) /Amulet device (St. Jude Medical, Minneapolis, Minnesota) was shown to be non-inferior but also superior as compared to warfarin in preventing the combined outcome of stroke, systemic embolism, and cardiovascular death. Therefore, LAAC has become an integral part of treatment guidelines in AF patients.

However, the post procedural management of antithrombotic therapy in these patients remains a challenge, as bleeding risk needs to be balanced against risk for thrombus formation on the device and thromboembolic complications. After LAAC, various antithrombotic protocols have been proposed by different teams but the optimal postprocedural antithrombotic medication and its duration are still debated. The Investigators recently showed in a prospective registry that LAAC using ACP devices followed by a single antiplatelet therapy could be a reasonable alternative for stroke prevention in patients with high bleeding risk.

The APPENDAGE study is a phase 4 multicentre randomized opened clinical trial comparing 2 different antithrombotic strategies (aspirin versus aspirin + clopidogrel) following LAAC. The primary objective of the study is to evaluate the efficacy of these 2 strategies after LAAC by comparing the occurrence of ischemic lesions on cerebrovascular MRI studies performed immediately after the procedure (D 0) and after 3 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with LAAC indication according to "Commission nationale d'évaluation des dispositifs médicaux et des technologies de santé" (CNEDiMTS) (National Commission for the Evaluation of Medical Devices and Health Technologies) guidelines
* Age ≥ 18 years
* Written informed consent provided by the patient
* Heart team approval: multidisciplinary team including interventional cardiologists, neurologists and other physicians discussing the definitive contraindication for anticoagulation
* Registration under social security system

Exclusion Criteria:

* Minors
* Unacceptable bleeding risk with double antiplatelet therapy decided by the physician who contraindicated oral anticoagulation
* LAAC contraindication : left appendage thrombus
* Major disease resulting in a life expectancy of < 1 year
* Severe and inherited bleeding disorder
* Known hypersensitivity to aspirin and/or clopidogrel:

  * Hypersensitivity to clopidogrel, acetylsalicylic acid, or one of the excipients or other nonsteroidal anti-inflammatory drugs (cross-reaction).
  * Asthma or a history of asthma with or without nasal polyps induced by salicylates or substances of close activity, including nonsteroidal anti-inflammatory drugs.
  * Evolving peptic ulcer or history of gastric hemorrhage or perforation after treatment with acetylsalicylic acid or other nonsteroidal anti-inflammatory drugs.
  * Any constitutional or acquired haemorrhagic disease.
  * Patients with mastocytosis, in whom the use of acetylsalicylic acid can lead to severe hypersensitivity reactions (including circulatory shocks with flushing, hypotension, tachycardia and vomiting).
  * Severe liver failure.
  * Severe kidney failure (Creatinine light < 30ml/min).
  * Uncontrolled severe heart failure
* Contraindication to MRI: claustrophobia or inability to lie still for exam time, implantable pacemaker or defibrillator, intracorporeal metal foreign body (especially intraocular), intracranial metal clip, cochlear implant, cardiac valve prosthesis type Starr-Edwards pre 6000, or biomedical device type insulin pump or neurostimulator.
* Guardianship
* Curatorship
* Pregnancy or child-bearing potential female
* Woman of childbearing age who does not benefit from highly effective contraception (CTFG recommendation on highly effective contraceptive methods: oral, intravaginal or transdermal estrogeno-progestin contraception; progestin-based oral, injectable or implantable contraception; intrauterine device; hormonal intrauterine device; female sterilization (occlusion of the fallopian tubes))
* Iode contraindication
* Patient already participating in another category 1 interventional research
* Patient in a period of exclusion relative to another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-05-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of ischaemic lesions number at 3 months appearing on brain MRI scans | Baseline and 3 months
  Assessment of number of ischaemic lesions appearing on diffusion sequences and/or (Fluid Attenuated Inversion Recovery) FLAIR between cerebral MRI scans at D0 after implantation and after 3 months of antithrombotic treatment. The interpretation of the MRI scans will be centralised and carried out by an independent Corelab in the neuro radiology imaging department of Bordeaux University Hospital. These analyses will be carried out by two independent radiologists. In the event of disagreements or inconsistent values, a third review will be carried out by a third independent radiologist. The final value of the different variables will be reduced to the average of these 2 or 3 interpretations.

SECONDARY OUTCOMES:
Occurrence of symptomatic cerebral ischaemic events | From day 1 to month 3
  Number of cerebral infarctions and transient ischaemic attacks identified by MRI and systematic neurological examination at D1 and M3, and at any time in the event of a symptomatic event.
Occurrence of systemic thromboembolic events | From day 1 to month 3
  Number of systemic thromboembolic events that will be identified when clinically symptomatic
Occurrence of cerebral haemorrhagic events | From day 0 to month 3
  Number of cerebral haemorrhagic events that will be identified by MRI and by systematic neurological examination at D0 and M3, and at any time in the event of a symptomatic event
Occurence of systemic bleeding events | From day 1 to month 3
  Number of systemic bleeding events that will be identified when clinically symptomatic
Assessment by the NIHSS scale (National Institute of Health Stroke Score) of the functional impact of ischaemic and/or haemorrhagic strokes | Day 1 and month 3
  It will be measured by the NIHSS scale score. Values range from 0 to 42. Score 1 to 4: minor stroke, 5 to 15 : moderate stroke, 15 to 20 : severe stroke, > 20 : severe stroke
Assessment by the Modified Rankin Score of the functional impact of ischaemic and/or haemorrhagic strokes | Day 1 and month 3
  It will be measured by the Modified Rankin Score. Values range from 0 (no symptoms) to 5 (severe disability)
Cognitive assessment by the Montreal Cognitive Assessment (MoCA) scale | Day 1 and Month 3
  Patients cognitive assessment will be performed using the Montreal Cognitive Assessment (MoCA) scale score. Values range from 0 to 30. A score of 26 is considered normal.
Occurrence of procedural related complications | From day 0 to month 3
  The number of procedural related complications (device embolization, significant pericardial effusion) will be assessed by physical examination and transthoracic echocardiography
Occurence of device-related thrombus, persistence of a residual leak and endothelialisation process | Month 3
  The number of device-related thrombus, persistence of a residual leak and endothelialisation process will be assessed by cardiac computed tomography (CT)
Counting of treatments taken | Month 3
  Compliance will be assessed for all patients by counting the number of treatments taken versus those that should have been taken. This compliance will be correlated with thromboembolic and hemorrhagic events to define the imputability of the therapeutic strategy on these events.

CONTACTS AND LOCATIONS:
Overall Officials: Zakaria JALAL, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Bordeaux University Hospital, Pessac
  - Toulouse University Hospital, Toulouse